CLINICAL TRIAL: NCT06961149
Title: Linked-Color Imaging Versus Indigo Carmine Pump Spraying on the Colorectal Adenoma Detection Rate: a Prospective , Randomized Controlled, Non-inferiority Study
Brief Title: Linked-Color Imaging Versus Indigo Carmine Pump Spraying on the Colorectal Adenoma Detection Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLL-202502-013-1
Record Dates: First submitted 2025-04-20; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Colonic Polyps; Adenomatous Polyps; Adenoma Detection Rate; Chromoendoscopy; Colorectal Neoplasms
Keywords: Adenoma Detection Rate; Linked-color imaging; Chromoendoscopy; Colonoscopy; Indigo Carmine
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linked-color imaging endoscopy (Experimental): Patients in this group will be carefully observed with LCI endoscopy during the colonoscopy withdraw.
  Interventions: Procedure: Linked-color imaging endoscopy
- Chromoendoscopy with indigo carmine solution spray (Active Comparator): Patients in this group will be carefully observed with spraying indigo carmine solution during the colonoscopy withdraw.
  Interventions: Procedure: Chromoendoscopy with indigo carmine solution spray

INTERVENTIONS:
Procedure: Chromoendoscopy with indigo carmine solution spray — Patients will undergo chromoendoscopy with spraying indigo carmine.
  Arms: Chromoendoscopy with indigo carmine solution spray
Procedure: Linked-color imaging endoscopy — Patients will undergo Linked-color imaging endoscopy.
  Arms: Linked-color imaging endoscopy

SUMMARY:
Detection and removal of polyps during colonoscopy is crucial for the prevention of colorectal cancer. Indigo carmine spraying up to the colonic mucosa could probably increase the adenoma detection rate, but considering the long withdrawal time of the endoscope and the resulting increase in time and cost. Linked-color imaging (LCI) is a newly developed image-enhanced endoscopy technology. It relies on wave length optimization of three colors (red, green, and blue) to make the lesions appear fuller. LCI improves the visibility of colorectal adenomas and polyps and may increase the detection rate of lesions. In order to explore the clinical application value of Linked-color imaging endoscopy, we performed a prospective, randomized controlled trial to compare adenoma detection rate of Linked-color imaging endoscopy and indigo carmine chromoendoscopy.

DETAILED DESCRIPTION:
If patients scheduled for colonoscopy meet the inclusion criteria but not the exclusion criteria, participants will be recruited to the study and randomized to one of two groups. Group allocation was revealed to endoscopists upon confirmation of cecal intubation. participants in Group A (treatment group) will undergo colonoscopy with LCI. participants in Group B (control group) will undergo spraying indigo carmine solution during withdrawal process. Any lesions found during the procedure will be removed and sent for pathological examination. The investigator will record the participants' general information (such as gender, age, symptoms, body mass index，etc.), colonoscopy data (such as duration etc.), and lesion characteristics (such as location, morphology, histopathological classification, etc.). All data were analyzed according to the ITT analysis, and the PP analysis was performed for all outcomes. Continuous variables were presented as means ± standard deviation (SD), and compared using Independent Samples t test. Categorical variables were expressed as frequency counts (percentages) and analyzed using Pearson's chi-square test or the Fisher exact test. Statistical analyses were performed using SPSS 27.0. Statistical significance was defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 45 and 85 years
2. Patients with a history of colorectal adenoma
3. Patients whose first-degree relatives have a history of colorectal cancer or colorectal adenoma
4. Patients with gastrointestinal symptoms (abdominal pain, bloody stool, chronic diarrhea or constipation, Unexplained anemia or weight loss;
5. Patients with positive Fecal Immunochemical Test

Exclusion Criteria:

1. Patients with pregnancy, inflammatory bowel disease, familial adenomatosis polyposis, suspected CRC; intestinal obstruction, coagulopathy
2. Patients with aspirin, clopidogrel or other anticoagulants/ antiplatelet drugs intake within 7 days
3. Patents previous colorectal resection
4. Patients with failed cecal intubation
5. Patients with inadequate bowel preparation quality (BBPS≤5)
6. Patients who refuse to participate or to provide informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate(ADR) | Periprocedural
  adenoma detection rate (ADR) defined as the percentage of patients with at least one histologically confirmed adenomatous polyp detected and resected during colonoscopy.

SECONDARY OUTCOMES:
detected rate of different lesions | Periprocedural
  detected rate of different lesions（advanced adenoma, sessile serrated lesion） adenoma per colonoscopy (APC) withdrawal time adverse event rates

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China